CLINICAL TRIAL: NCT01321294
Title: Laparoscopic Nissen Versus Toupet Fundoplication: Objective and Subjective Results of a Prospective Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Public Hospital Zell am See (Other)
Other Study IDs: Zell01
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Gastroesophageal Reflux Disease; Laparoscopic Antireflux Surgery
MeSH Terms: conditions — Gastroesophageal Reflux

ARMS (2):
- Nissen fundoplication (Active Comparator)
  Interventions: Procedure: laparoscopic anti-reflux surgery
- Toupet fundoplication (Active Comparator)
  Interventions: Procedure: laparoscopic anti-reflux surgery

INTERVENTIONS:
Procedure: laparoscopic anti-reflux surgery

SUMMARY:
The aim of this study is to compare subjective and objective outcome and surgical "side effects" of Nissen and Toupet fundoplication performed in a single institution by only two surgeons and to compare pre and postoperative findings to healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastroesophageal reflux disease
* Long history of GERD symptoms
* Persistent or recurrent symptoms despite optimal medical treatment
* Persistent or recurrent complications of GERD
* Reduced quality of life owing to increasing esophageal exposure to gastric juice
* Pathological values in the preoperative evaluated functional parameters

Exclusion Criteria:

* Previous esophageal or gastric surgery
* Poor physical status (American Society of Anesthesiologists (ASA) scores III and IV)
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- General Public Hospital Zell am See, Zell am See, Salzburg, Austria

REFERENCES:
- [Derived] Koch OO, Kaindlstorfer A, Antoniou SA, Luketina RR, Emmanuel K, Pointner R. Comparison of results from a randomized trial 1 year after laparoscopic Nissen and Toupet fundoplications. Surg Endosc. 2013 Jul;27(7):2383-90. doi: 10.1007/s00464-013-2803-0. Epub 2013 Jan 30. PMID 23361260